CLINICAL TRIAL: NCT05180149
Title: Personality and Drug Use (PDU)
Acronym: PDU
Status: Withdrawn | Type: Observational
Why Stopped: The sponsor of the study has changed. The study will be released, managed and registered by another institution who will be acting as a responsible party.
Sponsor: Quantified Citizen Technologies Inc. (Industry)
Collaborators: Maastricht University (Other); Psychedelic Data Society (Other)
Responsible Party: Principal Investigator, Maggie Kiraga, Research Associate, Maastricht University
Other Study IDs: QCPUBLICPDU1
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Personality
Keywords: Personality; Substance Use; Psychedelics; Drugs; Changes in Personality
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Psychedelics-only Group: A group of participants who reported using in their past psychedelic substances only (both classical and non-classical psychedelics are included). Specifically, in the current study this group included reports on the following substances:
  Psilocybin (magic mushrooms, truffles) LSD (acid) Mescaline (peyote, san pedro) Dimethyltryptamine (DMT) Ayahuasca 5-MeO-DMT 3-MMC Ibogaine Salvia Phenethylamines (2C family)
- Stimulants-only Group: A group of participants who reported using in their past drugs identified as stimulating compounds only (both recreational and prescribed usages are included). Stimulating compounds are considered, in the context of the current study, substances that increase the overall activity of the central nervous system. Specifically, in the current study this group included reports on the following substances:
  Cocaine Crack Amphetamines Methamphetamines Prescription stimulants (e.g., Adderall, Ritalin, Concerta)
- Depressants-only Group: A group of participants who reported using in their past drugs identified as depressing compounds only (both recreational and prescribed usages are included). Depressing compounds are considered, in the context of the current study, substances that decrease the overall activity of the central nervous system. Specifically, in the current study this group included reports on the following substances:
  Benzodiazepines Opiates (recreational use of heroin, opium, hydrocodone, oxycodone, oxymorphone, codeine, fentanyl) Prescription opioids
- Cannabinoids Group: A group of participants who reported using in their past cannabinoids compounds only (both recreational and prescribed usages are included). Specifically, in the current study this group included reports on the following substances:
  THC (cannabis, marijuana) CBD Medical Cannabis (both THC and CBD)
- Psychedelic and Non-psychedelic Substances Group: A group of participants who reported using in their past drugs identified as psychedelics and stimulants and/or depressants (both recreational and prescribed usages are included). In this group participants will be included who reported using at least one non-psychedelic drug additionally to a psychedelic one. Specifically, the following options were provided:
  1. Psychedelic compounds:
     Psilocybin (magic mushrooms, truffles) LSD (acid) Mescaline (peyote, san pedro) Dimethyltryptamine (DMT) Ayahuasca 5-MeO-DMT 3-MMC Ibogaine Salvia Phenethylamines (2C family)
  2. Non-psychedelic compounds:
  THC (cannabis, marijuana) Medical Cannabis (both THC and CBD) CBD MDMA (ecstasy) Ketamine Cocaine Crack Amphetamines Methamphetamines Prescription stimulants (e.g., Adderall, Ritalin, Concerta) Benzodiazepines Opiates (e.g., heroin, opium, hydrocodone, oxycodone, oxymorphone, codeine, fentanyl) Prescription opioids
- Substance-naive Group: A group of participants who reported no past experience with any of the substances listed in the current study nor reported using other substances (excluding alcohol and nicotine). Participants will be assigned to this group if and only if they choose the "None of the above" option from the Substance Use Survey (item 1).

SUMMARY:
The study aims to assess whether the use of drugs relates to personality ratings. Specifically, we plan to investigate if people with different histories of substance use differentiate on personality assessments (current and past).

DETAILED DESCRIPTION:
The study aims to assess the association between the use of various substances (including psychedelic and non-psychedelic drugs) and personality profiles. Specifically, the association between past drug usage and personality profiles will be investigated. As psychedelics were found to influence changes in personality over time, the present study aims to measure both the current personality profile (via the Big Five Inventory-44 (BFI)) and perceived retrospective changes in personality (via a self-constructed Retrospective Personality Scale (RPS)). To our knowledge, no study has explored the diversity of substance use histories in relation to individual current and retrospective personality traits and aggregate personality profiles.

This project aims to survey a large number of participants from all around the world, using a mobile app-based survey. The remote character of the study will increase its accessibility and diversity, which are common shortcomings in the psychedelic line of research. Additionally, a remote, anonymous study setup with no face-to-face interactions might help overcome any potential concerns participants may have regarding the sharing of sensitive information (e.g., reports on illicit substance use).

To increase scientific transparency and for educational purposes, the study team plans to share results summaries (comparisons of personalized results with the aggregated ones among participants sharing similar characteristics e.g., age, substance use history), which might be an additional motivating factor for study completion. Lastly, given that drug use in the natural environment (excluding laboratory/experimental setting) is characterized by large substance diversity and poly-drug use, we aim for a large sample size (with a minimum of 36 subjects per substance(s) category) to perform subgroup analyses. Therefore, this large-scale, low-budget, naturalistic, retrospective, observational study aims to shed light on the aforementioned gap in the literature and to lay a foundation of evidence for further (observational and experimental) research within the field.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* full legal and mental capacity
* access to a smartphone (iOS and Android) with internet

Exclusion Criteria:

* not fluent in English
* not able to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (age of 18 or above) of full mental and legal capacities.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Current Personality Profile | Single baseline measurement
  Raw scores on each of dimensions of the Big Five Inventory

SECONDARY OUTCOMES:
Changes in Personality Profile | Single baseline measurement
  Raw scores on the positive and negative dimensions of the self-constructed (for the study needs) Retrospective Personality Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kim PC Kuypers, PhD, Principal Investigator — Maastricht University

IPD SHARING:
Plan to Share IPD: Yes
The study will be pre-registered on the Open Science platform, where study details will be shared and regularly updated. This will be an open access project, meaning that all collected data and data analysis will be made available for all interested parties (via OSF platform). Additionally, we will share the individual summary reports with all participants who completed the study. The report will be accessible via a mobile app used to collect the study data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The raw data and clinical study report will be made available within 12 months from the end date of data collection.
Access Criteria: Open access

REFERENCES:
- [Background] Kiraga MK, Mason NL, Uthaug MV, van Oorsouw KIM, Toennes SW, Ramaekers JG, Kuypers KPC. Persisting Effects of Ayahuasca on Empathy, Creative Thinking, Decentering, Personality, and Well-Being. Front Pharmacol. 2021 Oct 1;12:721537. doi: 10.3389/fphar.2021.721537. eCollection 2021. PMID 34658861
- [Background] Bouso JC, Gonzalez D, Fondevila S, Cutchet M, Fernandez X, Ribeiro Barbosa PC, Alcazar-Corcoles MA, Araujo WS, Barbanoj MJ, Fabregas JM, Riba J. Personality, psychopathology, life attitudes and neuropsychological performance among ritual users of Ayahuasca: a longitudinal study. PLoS One. 2012;7(8):e42421. doi: 10.1371/journal.pone.0042421. Epub 2012 Aug 8. PMID 22905130
- [Background] Bouso JC, Palhano-Fontes F, Rodriguez-Fornells A, Ribeiro S, Sanches R, Crippa JA, Hallak JE, de Araujo DB, Riba J. Long-term use of psychedelic drugs is associated with differences in brain structure and personality in humans. Eur Neuropsychopharmacol. 2015 Apr;25(4):483-92. doi: 10.1016/j.euroneuro.2015.01.008. Epub 2015 Jan 16. PMID 25637267
- [Background] Williams MT, Davis AK, Xin Y, Sepeda ND, Grigas PC, Sinnott S, Haeny AM. People of color in North America report improvements in racial trauma and mental health symptoms following psychedelic experiences. Drugs (Abingdon Engl). 2021;28(3):215-226. doi: 10.1080/09687637.2020.1854688. Epub 2020 Dec 10. PMID 34349358
- [Background] Martins SS, Sampson L, Cerda M, Galea S. Worldwide Prevalence and Trends in Unintentional Drug Overdose: A Systematic Review of the Literature. Am J Public Health. 2015 Nov;105(11):e29-49. doi: 10.2105/AJPH.2015.302843. PMID 26451760
- [Background] Harm reduction: An approach to reducing risky health behaviours in adolescents. Paediatr Child Health. 2008 Jan;13(1):53-60. doi: 10.1093/pch/13.1.53. No abstract available. PMID 19119355
- See also: Culture and psychedelic psychotherapy: Ethnic and racial themes from three Black women therapists — https://akjournals.com/view/journals/2054/4/3/article-p125.xml